CLINICAL TRIAL: NCT05802810
Title: The Mass Balance Study of [14C]JT001 in Chinese Healthy Adult Male Subjects
Brief Title: The Mass Balance Study of [14C]JT001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Vinnerna Biosciences Co., Ltd. (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JT016-001-I
Record Dates: First submitted 2023-02-17; First posted 2023-04-07 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]JT001 (Experimental)
  Interventions: Drug: [14C]JT001

INTERVENTIONS:
Drug: [14C]JT001 — Subjects will receive approximately 300 mg/100 µCi of [14C]JT001 orally.

SUMMARY:
This study is a single center, single dose, non-randomized, open design clinical study.By quantitative analysis of the biological samples of subjects after oral administration of [14C]JT001, the data of human radioactive excretion rate and the main excretion pathway will be obtained. The main metabolites ,metabolic pathways and elimination pathways of JT001 will be identified.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males
2. Age: 18-45 years old
3. Body weight: Body mass index (BMI) is between 19.0 and 26.0 kg/m2 (including boundary values), and the body weight of the subject is not less than 50.0 kg;
4. Voluntarily sign informed consent;
5. Subjects were able to complete the trail according to protocol.

Exclusion Criteria:

1. Physical examination, vital signs, routine laboratory examination, imaging examination abnormal and clinically significant
2. The electrocardiogram was abnormal and was considered clinically significant by the investigators, or has a history of organic heart disease
3. Has hepatitis B (HBV) or hepatitis C (HCV) or HIV antibody and syphilis antibody positive;
4. Any drug that inhibits or induces the drug transporters P-gp and BCRP has been used within 30 days prior to the screening period
5. Any conditions that may affect drug absorption.
6. Previous antineoplastic therapy meets washout requirements.
7. Hemorrhoids or perianal disease with regular/ongoing blood in the stool, irritable bowel syndrome, inflammatory bowel disease
8. Habitual constipation or diarrhea.
9. Significant radioactive exposure within 1 year.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2023-03-18 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Total radioactive recovery | 1 month
  The percentage of radioactivity recovered from collected samples
cumulative excretion rate of total radioactive material in fecal matter | 1 month
  After oral administration of the drug, the subjects collected feces for 10 Days to obtain the excretion of accumulated radioactive substances in feces
Peak concentration（Cmax） | 1 month
  The highest plasma drug concentration that can be achieved after medication
time to peak（Tmax） | 1 month
  After a single dose, the time of peak blood concentration
elimination half life（t1/2） | 1 month
  the time it takes the blood to reduce the concentration of the drug to half
Major metabolites in human plasma, urine, and feces by liquid chromatography-mass spectrometry (LC-MS/MS) | 1 month
  The main metabolites in plasma, urine and fecal samples will be identified by liquid chromatography-mass spectrometry (LC-MS/MS)

SECONDARY OUTCOMES:
Adverse events (AEs) | 2 month
  Number of cases and incidence of adverse events(AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No